CLINICAL TRIAL: NCT00180323
Title: ACC - Atrial Contribution to CRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACC Version 1.1 11/09/2003
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Results first posted 2012-11-12 (Estimated); Last update posted 2021-02-11 (Actual); Status verified 2021-01

CONDITIONS: Dilated Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Dilated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Renewal CRT (CRT ICD) (Experimental): Single arm study only. All patients will undergo advanced echocardiographic examination pre-operative, pre-discharge after implantation and at 3 and 6-months follow-up. AV-delay optimization will be performed using aortic VTI (Velocity Time Integral) measured by continuous wave Doppler in a modified 4-chamber view. During optimisation aortic VTI will be measured at different heart rates reached by increasing atrial pacing 10, 20 and 30 beats above intrinsic heart rate (IHR).
  Interventions: Device: Renewal

INTERVENTIONS:
Device: Renewal — Renewal is a CRT-D device for cardiac resynchronization therapy

SUMMARY:
This prospective study will evaluate in patients, fulfilling implant criteria for Cardiac Resynchronisation Therapy (CRT) implant, the optimal atrial contribution to the resynchronised ventricles in the event of right atrial pacing.

DETAILED DESCRIPTION:
All patients will undergo advanced echocardiographic examination pre-operative, pre-discharge after implantation and at 3 and 6-months follow-up. AV-delay optimization will be performed using aortic VTI measured by continuous wave Doppler in a modified 4-chamber view. During optimisation aortic VTI will be measured at different heart rates reached by increasing atrial pacing 10, 20 and 30 beats above intrinsic heart rate (IHR).

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of heart failure
* Left ventricular dysfunction
* Ventricular dyssynchrony
* 18 years or of legal age in order to give informed consent according to national laws
* Able to understand the nature of the procedure
* Available for follow-up on a regular basis at an approved investigational center

Exclusion Criteria:

* Atrial Fibrillation
* Life expectancy of less than six months due to other medical conditions
* For women: pregnancy or absence of medically accepted birth control
* Inability or refusal to sign the Patient Informed Consent
* Inability or refusal to comply with the follow up schedule or protocol requirements
* Inability to undergo device implant, including general anaesthesia if required
* Mechanical tricuspid prosthesis
* Currently enrolled in another investigational study, including drug investigations
* Hypertrophic Obstructive Cardiomyopathy (HOCM)
* Not meeting the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2004-11; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jasper Hastrup Svendson, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1
Started | 43
Completed | 43
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Group 1
Number analyzed (Participants) | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 31
Region of Enrollment [Number; unit: participants]
  Denmark | 43

OUTCOME MEASURES:

1. Primary Outcome: Aortic Velocity Time Integral (VTI)
Description: Velocity time integral of the aortic flow correlates with cardiac output and is an accepted parameter for optimization of Cardiac Resynchronization Therapy (CRT).
Time Frame: At implant (baseline), 3 months and 6 months Follow-up
Measure: Mean (Standard Deviation); unit: cm
Groups:
- Cardiac Resynchronization Therapy ICD (Renewal CRT): Velocity time integral will be measured at implant (baseline), 3 months and 6 months Follow-up. Measurements will be taken at each timepoint at intrinsic heart rate and 10, 20 and 30 Bpm above intrinsic heart rate (paced rhythm)
Arm/Group | Cardiac Resynchronization Therapy ICD (Renewal CRT)
Number analyzed (Participants) | 43
cm
  VTI at baseline intrinsic rhythm | 22.4 (7.7)
  VTI at baseline intrinsic rhythm + 10 Bpm | 21.7 (7.7)
  VTI at baseline intrinsic rhythm + 20 Bpm | 19.4 (7.5)
  VTI at baseline intrinsic rhythm + 30 Bpm | 18.1 (7.1)
  VTI at 3M Follow-up intrinsic rhythm | 23.6 (9.0)
  VTI at 3M Follow-up intrinsic rhythm + 10 Bpm | 21.9 (9.0)
  VTI at 3M Follow-up intrinsic rhythm + 20 Bpm | 21.2 (8.1)
  VTI at 3M Follow-up intrinsic rhythm + 30 Bpm | 19.4 (8.3)
  VTI at 6M Follow-up intrinsic rhythm | 24.6 (8.4)
  VTI at 6M Follow-up intrinsic rhythm + 10 Bpm | 23.2 (7.5)
  VTI at 6M Follow-up intrinsic rhythm + 20 Bpm | 21.7 (7.0)
  VTI at 6M Follow-up intrinsic rhythm + 30 Bpm | 20.2 (7.2)

2. Primary Outcome: Optimal AV-Delay (AVD)
Description: Optimal AV-Delay will be measured at implant (baseline ), 3months and 6 months Follow-up for intrinsic heart rate, and 10, 20 and 30 Bpm above intrinsic heart rate.
Time Frame: Implant (baseline), 3 months and 6 months Follow-up
Measure: Mean (Standard Deviation); unit: ms
Groups:
- Cardiac Resynchronization Therapy ICD (Renewal CRT): Optimal AV-Delay will be measured at implant (baseline ), 3months and 6 months Follow-up for intrinsic heart rate, and 10, 20 and 30 Bpm above intrinsic heart rate.
Arm/Group | Cardiac Resynchronization Therapy ICD (Renewal CRT)
Number analyzed (Participants) | 43
ms
  Optimal AVD at baseline intrinsic rhythm | 115 (24)
  Optimal AVD at baseline intrinsic rhythm +10Bpm | 119 (29)
  Optimal AVD at baseline intrinsic rhythm +20Bpm | 123 (22)
  Optimal AVD at baseline intrinsic rhythm +30Bpm | 127 (28)
  Optimal AVD at 3M intrinsic rhythm | 117 (28)
  Optimal AVD at 3M intrinsic rhythm +10Bpm | 117 (24)
  Optimal AVD at 3M intrinsic rhythm +20Bpm | 127 (28)
  Optimal AVD at 3M intrinsic rhythm +3Bpm | 119 (23)
  Optimal AVD at 6M intrinsic rhythm | 115 (24)
  Optimal AVD at 6M intrinsic rhythm +10Bpm | 132 (28)
  Optimal AVD at 6M intrinsic rhythm +20Bpm | 130 (30)
  Optimal AVD at 6M intrinsic rhythm +30Bpm | 130 (17)

3. Secondary Outcome: 6 Minute Walk Test
Description: 6 Minute Walk Test was performed at implant (baseline), 3 months and 6 months follow-up Distance walked within 6 minutes is assessed in meter. This is a test that reflects daily life activities of elderly patients.
Time Frame: implant (baseline), 3 months and 6 months Follow-up
Measure: Mean (Standard Error); unit: meter
Groups:
- Cardiac Resynchronization Therapy ICD (Renewal CRT): 6 minute walktest (6 MWT) was performed before implant (baseline ), 3months and 6 months Follow-up.
Arm/Group | Cardiac Resynchronization Therapy ICD (Renewal CRT)
Number analyzed (Participants) | 43
meter
  6 MWT at baseline | 388 (88)
  6 MWT at 3M Follow-up | 470 (87)
  6 MWT at 6M Follow-up | 497 (83)

4. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF)
Description: Left ventricular Ejection Fraction (LVEF) was measured before implant (baseline) and at 3 and 6 months Follow-up
Time Frame: implant (baseline), 3 Months, 6 Months
Measure: Mean (Standard Deviation); unit: % of cardiac volume
Arm/Group | Cardiac Resynchronization Therapy ICD (Renewal CRT)
Number analyzed (Participants) | 43
% of cardiac volume
  LVEF at baseline | 21 (6)
  LVEF at 3M | 24 (7)
  LVEF at 6M | 24 (8)

ADVERSE EVENTS:
Time Frame: Adverse events were assessed only at implant, 3 months and 6 months follow-up. Events observed between these visits were not provided by the investigator.
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 0/43
Other Adverse Events (participants affected / at risk) | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No